CLINICAL TRIAL: NCT00039793
Title: Massage Therapy for Cancer-Related Fatigue
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R21AT000348-01 (NIH); NCT00058513 (obsolete NCT alias)
Record Dates: First submitted 2002-06-11; First posted 2002-06-13 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-07

CONDITIONS: Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms
Keywords: Cancer-related fatigue; alternative medicine; cancer rehabilitation /care; fatigue; human therapy evaluation; physical therapy; neoplasm /cancer chemotherapy; neoplasm /cancer palliative treatment
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Colorectal Neoplasms; Fatigue

INTERVENTIONS:
Procedure: Moderate-intensity and low-intensity bodywork therapy

SUMMARY:
The purpose of this study is to develop methods for studying the effect of bodywork therapy on symptoms of fatigue in patients undergoing cancer chemotherapy.

DETAILED DESCRIPTION:
The proposed project is a randomized pilot trial of a Swedish-style massage therapy intervention for the treatment of fatigue in patients who are undergoing cancer chemotherapy. Fatigue is the most common complaint of patients receiving treatment for cancer, but is often difficult to treat and causes a substantial decrement in patients' quality of life. Massage therapy is a non-invasive intervention used in many patients with cancer for symptom control. Prior small studies have suggested some efficacy of bodywork therapies in conditions characterized by fatigue, such as fibromyalgia and chronic fatigue syndrome. Based on these results, massage therapy may provide an important adjunct in ameliorating fatigue and enhancing cancer patients' well being.

The proposed study is a 12-week, randomized, three-arm, parallel-comparison clinical trial comparing the effects of a Swedish-style massage regimen to a sham bodywork control and a usual-care group for fatigue reduction in cancer patents undergoing chemotherapy. Patients with breast, ovarian, prostate, or colo-rectal cancer will be enrolled; the primary outcome measure is a quantitative assessment of fatigue symptoms. This study will determine efficacy, functioning, perceptions of fatigue, and quality of life. This study should provide not only important data on the potential efficacy of massage therapy for the treatment of fatigue, but also advance the methodology for studying CAM interventions for difficult-to-treat symptomatic conditions.

ELIGIBILITY:
Inclusion criteria:

* Confirmed tissue diagnosis of cancer of the breast, ovary, prostate or colo-rectum
* Have an anticipated completion of chemotherapy no more than 2 weeks before the last bodywork session.
* Have a primary oncologist
* Currently receiving chemotherapy or completed chemotherapy treatment within the past 6 months

Exclusion criteria:

* Active skin rash or open cutaneous lesions.
* History of venous thrombosis (or symptomatic varicosity)
* Identification of a thrombosis using an ultrasound test of the legs.
* Long term (> 3 months) steroid medications for other medical conditions in past 5 years
* Plans to move out of the study region within 6 months
* Thyroid-stimulating hormone (TSH) level above the upper limit of normal
* Hematocrit <25%
* Platelet count of < 50,000
* Patients who have been receiving regular (i.e. at least twice a month) bodywork over the past 6 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Start 2001-03; Study Completion 2004-03

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Avins, MD, MPH, Principal Investigator — Osher Center for Integrative Medicine, University of California, San Francisco; Shelley Adler, PhD — Osher Center for Integrative Medicine, University of California, San Francisco; Michael Patterson, MS — Osher Center for Integrative Medicine, University of California, San Francisco
Locations (1):
- Osher Center for Integrative Medicine, San Francisco, California, United States

REFERENCES:
- [Derived] Patterson M, Maurer S, Adler SR, Avins AL. A novel clinical-trial design for the study of massage therapy. Complement Ther Med. 2008 Jun;16(3):169-76. doi: 10.1016/j.ctim.2007.08.001. Epub 2007 Sep 21. PMID 18534330
- See also: Click here for more information about how to contact this study — http://www.ucsf.edu/ocim/